CLINICAL TRIAL: NCT01556594
Title: Phase II Study to Investigate the Safety and Efficacy of 2 Dose Levels of a Novel Glucagon Formulation Compared to Commercially Available Glucagon in Type 1 Diabetic Patients Following Insulin-induced Hypoglycemia
Brief Title: Safety and Efficacy of a Novel Glucagon Formulation in Type 1 Diabetic Patients Following Insulin-induced Hypoglycemia
Acronym: AMG102
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Locemia Solutions ULC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 16416; I8R-MC-IGBA (Other: Eli Lilly and Company); AMG102 (Other: Locemia Solutions ULC)
Record Dates: First submitted 2012-03-15; First posted 2012-03-16 (Estimated); Results first posted 2014-08-13 (Estimated); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Hypoglycemia
Keywords: Hypoglycemia; Diabetes mellitus
MeSH Terms: conditions — Hypoglycemia; Diabetes Mellitus | interventions — Glucagon; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Nasal Glucagon 1 mg (Experimental): Nasal glucagon (NG) administered as single dose of 1 milligram (mg).
  Interventions: Drug: Nasal Glucagon 1 mg
- Nasal Glucagon 2 mg (Experimental): NG administered as single dose of 2 mg.
  Interventions: Drug: Nasal Glucagon 2 mg
- SC Glucagon (Active Comparator): Glucagon solution dose of 1 mg administered as a single subcutaneous (SC) injection.
  Interventions: Drug: SC Glucagon
- Nasal Glucagon 3 mg (Experimental): NG administered as single dose of 3 mg (composed of one dose of 1 mg NG immediately followed by one dose of 2mg NG).
  Interventions: Drug: Nasal Glucagon 3 mg

INTERVENTIONS:
Drug: Nasal Glucagon 1 mg
  Other Names: Dry Powder Nasal Glucagon; AMG504-1; LY900018
  Arms: Nasal Glucagon 1 mg
Drug: Nasal Glucagon 2 mg
  Other Names: Dry Powder Nasal Glucagon; AMG504-1; LY900018
  Arms: Nasal Glucagon 2 mg
Drug: SC Glucagon
  Other Names: Glucagon; Glucagon for injection (rDNA origin)
  Arms: SC Glucagon
Drug: Nasal Glucagon 3 mg
  Other Names: Dry Powder Nasal Glucagon; AMG504-1; LY900018
  Arms: Nasal Glucagon 3 mg

SUMMARY:
In this study, participants with Type 1 diabetes received insulin through an infusion into a vein to reduce their blood glucose, and then received nasal glucagon (NG) or glucagon for injection under the skin, and their blood glucose was measured for 3 hours.

The main objective of this study was to evaluate the safety and efficacy of intranasal and subcutaneous glucagon (SC) in reversing insulin-induced hypoglycemia in participants with type 1 diabetes.

DETAILED DESCRIPTION:
In the study, up to four (4) treatments were administered as a single dose either intranasally or subcutaneously to eighteen (18) male or female participants under fasting conditions and following the use of insulin to lower blood glucose. The participants were assigned at random to a group that received one treatment for each of the 3 study periods. The glucagon administrations were separated by approximately 7 calendar days. For 2 participants, a single dose of 3 mg NG was administered at the 4th period that was separated by at least 21 calendar days from the 3rd period.

ELIGIBILITY:
Inclusion Criteria:

* History of type 1 diabetes between 2 and 30 years
* Receiving daily insulin injections or insulin pump therapy for at least 2 years
* If patient is taking Lantus, Levemir or equivalent once-daily in the evening as basal insulin, must be willing to transition to once-daily in the morning at least 48 hours prior to 1st dosing, and to follow this dosing regimen for the entire duration of the study
* Body mass index (BMI) greater than or equal to 20.00 and below or equal to 33.00 kg/m2
* Female patients must not be pregnant, and must be using effective contraception.
* Light-, non- or ex-smokers. A light smoker is defined as someone smoking 10 cigarettes or less per day for at least 3 months before day 1 of this study. An ex smoker is defined as someone who completely stopped smoking for at least 6 months before day 1 of this study

Exclusion Criteria:

* History of an episode of severe hypoglycemia (as defined by an episode that required third party assistance for treatment) in the previous 6 months before day 1 of this study
* Score ≥4 on the Clarke Hypoglycemia Awareness survey at screening
* Presence or history of pheochromocytoma (i.e. adrenal gland tumor)
* Presence or history of significant upper respiratory or allergic (i.e., seasonal rhinitis) disease
* Presence of clinically significant findings on nasal examination and bilateral anterior rhinoscopy
* Known presence of hereditary problems of galactose and /or lactose intolerance
* History of significant hypersensitivity to glucagon or any related products as well as severe hypersensitivity reactions (like angioedema) to any drugs

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2012-03; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Algorithme Pharma, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the clinical site's database and from participants who responded to advertising in local media.
Groups:
- Treatment Group 1: Nasal glucagon (NG) dose of 1 milligram (mg) and 2 mg. Subcutaneous (SC) glucagon dose of 1mg.
- Treatment Group 2: NG dose of 1 mg, 2 mg and 3mg. SC glucagon dose of 1mg.
- Treatment Group 3: NG dose of 2 mg and 3mg. SC glucagon dose of 1mg.
Period: Overall Study
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3
Started | 10 | 2 | 6
Completed | 10 | 2 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Treatment Group 1: NG dose of 1 mg and 2 mg. SC glucagon dose of 1mg.
- Total: Total of all reporting groups
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Total
Number analyzed (Participants) | 10 | 2 | 6 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 2 | 6 | 18
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (14) | 42 (2) | 25 (6) | 32 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 0 | 1 | 5
  Male | 6 | 2 | 5 | 13
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 10 | 2 | 6 | 18

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Responders
Description: Participants with a blood glucose increment of ≥1.5 millimole per liter [mmol/L) within 15 of nadir (5 minutes post dose) and for at least 10 minutes following nadir.
Time Frame: Pre-dose; 30 minutes following glucagon administration
Population: All enrolled participants.
Measure: Number; unit: percentage of participants
Groups:
- SC Glucagon: SC glucagon injection 1 mg
- NG 1 mg: NG dose of 1 mg
- NG 2 mg: NG dose of 2 mg
- NG 3 mg: NG dose of 3 mg
Arm/Group | SC Glucagon | NG 1 mg | NG 2 mg | NG 3 mg
Number analyzed (Participants) | 18 | 12 | 18 | 8
percentage of participants | 83.3 | 25 | 50 | 75

2. Primary Outcome: Number of Participants With at Least One Adverse Event
Description: Safety and tolerability evaluated through the assessment of adverse events. An AE was defined as any untoward medical occurrence in a clinical investigation subject administered the investigational product and which did not necessarily have a causal relationship with this treatment. A summary of other nonserious AEs, and all SAE's, regardless of causality, is located in the Reported Adverse Events section.
Time Frame: Within 3 hours post glucagon administration
Population: Participants who received at least one dose of glucagon (SC Glucagon or NG).
Measure: Count of Participants; unit: Participants
Arm/Group | SC Glucagon | NG 1 mg | NG 2 mg | NG 3 mg
Number analyzed (Participants) | 18 | 12 | 18 | 8
Participants | 16 | 9 | 15 | 8

3. Secondary Outcome: Maximum Concentration (Cmax) of Baseline-Adjusted Glucose
Time Frame: Pre-dose; 0.08, 0.17, 0.25, 0.33, 0.5, 0.67, 1.0, 1.5, 2.0, 2.5 and 3.0 hours after glucagon administration
Population: Participants who received at least one dose of glucagon (SC Glucagon or NG).
Measure: Mean (Standard Deviation); unit: millimole per liter (mmol/L)
Arm/Group | SC Glucagon | NG 1 mg | NG 2 mg | NG 3 mg
Number analyzed (Participants) | 18 | 9 | 17 | 8
millimole per liter (mmol/L) | 5.68 (2.57) | 2.41 (1.89) | 3.46 (1.44) | 3.11 (2.08)

4. Secondary Outcome: Time to Maximum Concentration (Tmax) of Baseline-Adjusted Glucose
Time Frame: Pre-dose; 0.08, 0.17, 0.25, 0.33, 0.5, 0.67, 1.0, 1.5, 2.0, 2.5 and 3.0 hours after glucagon administration
Population: Participants who received at least one dose of glucagon (SC Glucagon or NG).
Measure: Median (Full Range); unit: hours (hr)
Arm/Group | SC Glucagon | NG 1 mg | NG 2 mg | NG 3 mg
Number analyzed (Participants) | 18 | 9 | 17 | 8
hours (hr) | 1.5 [0.5 to 3.0] | 0.67 [0.08 to 3.0] | 1.0 [0.5 to 3.0] | 1.0 [0.5 to 3.0]

5. Secondary Outcome: Maximum Change From Baseline Concentration (Cmax) of Glucagon
Time Frame: Pre-dose; 0.08, 0.17, 0.25, 0.33, 0.5, 0.67, 1.0, 1.5, 2.0, 2.5 and 3.0 hours after glucagon administration
Population: Participants who received at least one dose of glucagon (SC Glucagon or NG) with available pharmacokinetic data.
Measure: Mean (Standard Deviation); unit: picograms per millilitre (pg/mL)
Arm/Group | SC Glucagon | NG 1 mg | NG 2 mg | NG 3 mg
Number analyzed (Participants) | 18 | 5 | 14 | 8
picograms per millilitre (pg/mL) | 3930 (2650) | 504 (342) | 2370 (1810) | 1360 (722)

6. Secondary Outcome: Time to Maximum Concentration (Tmax) of Baseline Adjusted Glucagon
Time Frame: Pre-dose; 0.08, 0.17, 0.25, 0.33, 0.5, 0.67, 1.0, 1.5, 2.0, 2.5 and 3.0 hours after glucagon administration
Population: Participants who received at least one dose of glucagon (SC Glucagon or NG) with available pharmacokinetic data.
Measure: Median (Full Range); unit: hours (hr)
Arm/Group | SC Glucagon | NG 1 mg | NG 2 mg | NG 3 mg
Number analyzed (Participants) | 18 | 5 | 14 | 8
hours (hr) | 0.33 [0.08 to 0.67] | 0.25 [0.17 to 0.25] | 0.33 [0.17 to 0.50] | 0.29 [0.17 to 0.50]

7. Secondary Outcome: Area Under the Curve (AUC0-last) of Baseline Adjusted Glucagon
Time Frame: Pre-dose; 0.08, 0.17, 0.25, 0.33, 0.5, 0.67, 1.0, 1.5, 2.0, 2.5 and 3.0 hours after glucagon administration
Population: Participants who received at least one dose of glucagon (SC Glucagon or NG) with available pharmacokinetic data.
Measure: Mean (Standard Deviation); unit: hour*picogram per millilitre (hr*pg/mL)
Arm/Group | SC Glucagon | NG 1 mg | NG 2 mg | NG 3 mg
Number analyzed (Participants) | 18 | 5 | 14 | 8
hour*picogram per millilitre (hr*pg/mL) | 2390 (1350) | 95.2 (38.4) | 886 (796) | 720 (386)

ADVERSE EVENTS:
Time Frame: First dose of study drug (Day 1) until post-study completion (Day 38)
Description: All enrolled participants who received at least one dose of glucagon (SC Glucagon or NG).
Arm/Group | SC Glucagon | NG 1 mg | NG 2 mg | NG 3 mg
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/12 | 0/18 | 0/8
Other Adverse Events (participants affected / at risk) | 16/18 | 9/12 | 15/18 | 8/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SC Glucagon (N=18) | NG 1 mg (N=12) | NG 2 mg (N=18) | NG 3 mg (N=8)
Nausea (Gastrointestinal disorders) | 7 (7) | 1 (1) | 3 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (8) | 0 (0) | 0 (0) | 0 (0)
Lacrimation Increased (Eye disorders) | 1 (1) | 1 (1) | 9 (9) | 6 (7)
Eye pruritus (Eye disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 1 (1) | 6 (7) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 4 (5) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Feeling hot (General disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Asthenia (General disorders) | 2 (3) | 2 (3) | 5 (6) | 1 (1)
Hot flush (Vascular disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Pallor (Vascular disorders) | 4 (4) | 0 (0) | 2 (2) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Disturbance in attention (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 5 (5) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (4) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (2) | 0 (0)
Ear pruritus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ocular Hyperaemia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheter Site Bruise (General disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Catheter Site Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hunger (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vessel Puncture Site Bruise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal Dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal Pruritus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cold Sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No